CLINICAL TRIAL: NCT03895554
Title: Quantification of Myocardial Blood Flow by Positron Emission Tomography in Healthy Volunteers
Acronym: PET Normals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Robert Bober, M.D., Director of Cardiac Molecular Imaging, Ochsner Health System
Other Study IDs: STUDY00000188
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Normal Healthy Volunteers Without Chronic Medical Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Normal volunteers: Normal, healthy volunteers with undergo cardiac PET stress testing.
  Interventions: Procedure: cardiac PET stress test

INTERVENTIONS:
Procedure: cardiac PET stress test — Volunteers will undergo cardiac PET stress testing

SUMMARY:
To establish quantitative values of myocardial blood flow (MBF) in normal, healthy volunteers .

DETAILED DESCRIPTION:
We seek to establish quantitative values of myocardial blood flow in 20 normal, healthy volunteers using our existing 2D PET camera (Positron Attrius) and invasively validated software package (HeartSee) in order to 1) establish institutional values for which clinical patients can be compared to and 2) add to the collective data of the scientific community. Values to be measured will be resting myocardial blood flow (MBF), stress MBF and coronary flow reserve.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 and <40 years old
* Participants must be able to give informed consent.
* Ability to abstain from caffeine for 48 hours

Exclusion Criteria:

* Any chronic cardiac disease or condition (e.g. hypertension, hyperlipidemia)
* Any chronic systemic disease or condition (e.g. diabetes, systemic lupus, rheumatoid arthritis)
* Tobacco use
* Family history in a first degree relative with clinical coronary artery disease (history of myocardial infarctio, percutaneous intervention or coronary artery bypass grafting) in men <55 years old or women <65 years old
* Severe claustrophobia
* Positive urine pregnancy test
* Inability to give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers will be selected from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Absolute myocardial blood flow at rest and stress in cc/min/g | measured at the time of the cardiac PET stress scan
  resting and stress MBF are in units of cc/min/g

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Intention to publish the data in peer reviewed journal.

REFERENCES:
- [Background] Araujo LI, Lammertsma AA, Rhodes CG, McFalls EO, Iida H, Rechavia E, Galassi A, De Silva R, Jones T, Maseri A. Noninvasive quantification of regional myocardial blood flow in coronary artery disease with oxygen-15-labeled carbon dioxide inhalation and positron emission tomography. Circulation. 1991 Mar;83(3):875-85. doi: 10.1161/01.cir.83.3.875. PMID 1900224
- [Background] Bergmann SR, Herrero P, Markham J, Weinheimer CJ, Walsh MN. Noninvasive quantitation of myocardial blood flow in human subjects with oxygen-15-labeled water and positron emission tomography. J Am Coll Cardiol. 1989 Sep;14(3):639-52. doi: 10.1016/0735-1097(89)90105-8. PMID 2788669
- [Background] Sdringola S, Johnson NP, Kirkeeide RL, Cid E, Gould KL. Impact of unexpected factors on quantitative myocardial perfusion and coronary flow reserve in young, asymptomatic volunteers. JACC Cardiovasc Imaging. 2011 Apr;4(4):402-12. doi: 10.1016/j.jcmg.2011.02.008. PMID 21492816
- [Background] Renaud JM, DaSilva JN, Beanlands RS, DeKemp RA. Characterizing the normal range of myocardial blood flow with (8)(2)rubidium and (1)(3)N-ammonia PET imaging. J Nucl Cardiol. 2013 Aug;20(4):578-91. doi: 10.1007/s12350-013-9721-3. Epub 2013 May 9. PMID 23657833
- [Background] Merlet P, Mazoyer B, Hittinger L, Valette H, Saal JP, Bendriem B, Crozatier B, Castaigne A, Syrota A, Rande JL. Assessment of coronary reserve in man: comparison between positron emission tomography with oxygen-15-labeled water and intracoronary Doppler technique. J Nucl Med. 1993 Nov;34(11):1899-904. PMID 8229231
- [Background] Kern MJ, Bach RG, Mechem CJ, Caracciolo EA, Aguirre FV, Miller LW, Donohue TJ. Variations in normal coronary vasodilatory reserve stratified by artery, gender, heart transplantation and coronary artery disease. J Am Coll Cardiol. 1996 Nov 1;28(5):1154-60. doi: 10.1016/S0735-1097(96)00327-0. PMID 8890809
- [Background] Renaud JM, Yip K, Guimond J, Trottier M, Pibarot P, Turcotte E, Maguire C, Lalonde L, Gulenchyn K, Farncombe T, Wisenberg G, Moody J, Lee B, Port SC, Turkington TG, Beanlands RS, deKemp RA. Characterization of 3-Dimensional PET Systems for Accurate Quantification of Myocardial Blood Flow. J Nucl Med. 2017 Jan;58(1):103-109. doi: 10.2967/jnumed.116.174565. Epub 2016 Aug 18. PMID 27539843
- [Background] Gould KL, Johnson NP, Bateman TM, Beanlands RS, Bengel FM, Bober R, Camici PG, Cerqueira MD, Chow BJW, Di Carli MF, Dorbala S, Gewirtz H, Gropler RJ, Kaufmann PA, Knaapen P, Knuuti J, Merhige ME, Rentrop KP, Ruddy TD, Schelbert HR, Schindler TH, Schwaiger M, Sdringola S, Vitarello J, Williams KA Sr, Gordon D, Dilsizian V, Narula J. Anatomic versus physiologic assessment of coronary artery disease. Role of coronary flow reserve, fractional flow reserve, and positron emission tomography imaging in revascularization decision-making. J Am Coll Cardiol. 2013 Oct 29;62(18):1639-1653. doi: 10.1016/j.jacc.2013.07.076. Epub 2013 Aug 28. PMID 23954338
- [Background] Nesterov SV, Deshayes E, Sciagra R, Settimo L, Declerck JM, Pan XB, Yoshinaga K, Katoh C, Slomka PJ, Germano G, Han C, Aalto V, Alessio AM, Ficaro EP, Lee BC, Nekolla SG, Gwet KL, deKemp RA, Klein R, Dickson J, Case JA, Bateman T, Prior JO, Knuuti JM. Quantification of myocardial blood flow in absolute terms using (82)Rb PET imaging: the RUBY-10 Study. JACC Cardiovasc Imaging. 2014 Nov;7(11):1119-1127. doi: 10.1016/j.jcmg.2014.08.003. Epub 2014 Oct 8. PMID 25306543